CLINICAL TRIAL: NCT00881140
Title: The Effect of Vaginal Mifepristone on Reduction of Uterine Fibroids Size and the Symptoms Associated With the Fibroids - Pilot Study (Phase IIa)
Brief Title: Efficacy Study of Vaginal Mifepristone to Treat Uterine Fibroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioPro Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: bp001; 5300/08
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Uterine Fibroid; Vaginal Bleeding.
Keywords: oral mifepristone; vaginal tablets
MeSH Terms: conditions — Leiomyoma; Uterine Hemorrhage | interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- antiprogestin (Experimental): Daily use of 10 mg administrated per vagina
  Interventions: Drug: mifepristone vaginal tablets

INTERVENTIONS:
Drug: mifepristone vaginal tablets — Daily use of 10 mg administrated per vagina for 3 months
  Other Names: mifepristone

SUMMARY:
The purpose of this study is to evaluate the effect of daily dosage of vaginally mifepristone on reduction of uterine fibroids size and the symptoms associated with uterine fibroids.

DETAILED DESCRIPTION:
Uterine fibroids are benign tumors of the uterus made up of smooth muscle and the extracellular matrix proteins Collagen and Elastin. They are exceptionally common; the cumulative incidence of a diagnosis of fibroids in women aged 25 to 45 is approximately 30 percent.

Uterine fibroids can cause abnormal uterine bleeding, dysmenorrhea, lower back pain and non-cyclic pelvic pain. They also can contribute to symptoms related to an enlarging pelvic mass (e.g., urinary frequency or constipation).

Uterine fibroids are also associated with an increased risk of complications of pregnancy, and with infertility, although it is unclear whether this association is causative. Symptoms associated with uterine fibroids can have a significant impact on quality of life, with scores on standard measures that are comparable to those for other major chronic diseases

ELIGIBILITY:
Inclusion Criteria:

* Uninterested in fertility during the study.
* Premenopausal status.
* Active symptoms related to uterine fibroids.
* Subjects will be obligated to use non hormonal contraceptives during the study.

Exclusion Criteria:

* Abnormal liver and renal function
* Participants with significant increase in uterine fibroids size during a short time.
* Exclusionary health problems contraindicating mifepristone included adrenal disease; sickle cell anemia; severe liver, respiratory, or renal disease; and blood clotting defect.
* Current use of steroids, anticoagulants, herbals, or botanicals with possible hormonal effects.

Ages: 30 Years to 53 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Decrease of uterine fibroids volume by 25% and up. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Seidman, Prof', Principal Investigator — unaffiliation
Locations (2):
- Israel (2):
  - Rabin Medical Center, Petah Tikva, Hasaron
  - Gynecolaoy department - Shiba Medical Center Tel Hashomer, Ramat Gan

REFERENCES:
- [Background] Fiscella K, Eisinger SH, Meldrum S, Feng C, Fisher SG, Guzick DS. Effect of mifepristone for symptomatic leiomyomata on quality of life and uterine size: a randomized controlled trial. Obstet Gynecol. 2006 Dec;108(6):1381-7. doi: 10.1097/01.AOG.0000243776.23391.7b. PMID 17138770
- [Background] Steinauer J, Pritts EA, Jackson R, Jacoby AF. Systematic review of mifepristone for the treatment of uterine leiomyomata. Obstet Gynecol. 2004 Jun;103(6):1331-6. doi: 10.1097/01.AOG.0000127622.63269.8b. PMID 15172874
- [Background] Eisinger SH, Meldrum S, Fiscella K, le Roux HD, Guzick DS. Low-dose mifepristone for uterine leiomyomata. Obstet Gynecol. 2003 Feb;101(2):243-50. doi: 10.1016/s0029-7844(02)02511-5. PMID 12576246
- [Background] Spies JB, Coyne K, Guaou Guaou N, Boyle D, Skyrnarz-Murphy K, Gonzalves SM. The UFS-QOL, a new disease-specific symptom and health-related quality of life questionnaire for leiomyomata. Obstet Gynecol. 2002 Feb;99(2):290-300. doi: 10.1016/s0029-7844(01)01702-1. PMID 11814511
- [Background] Eisinger SH, Bonfiglio T, Fiscella K, Meldrum S, Guzick DS. Twelve-month safety and efficacy of low-dose mifepristone for uterine myomas. J Minim Invasive Gynecol. 2005 May-Jun;12(3):227-33. doi: 10.1016/j.jmig.2005.01.022. PMID 15922980
- [Background] Murphy AA, Kettel LM, Morales AJ, Roberts VJ, Yen SS. Regression of uterine leiomyomata in response to the antiprogesterone RU 486. J Clin Endocrinol Metab. 1993 Feb;76(2):513-7. doi: 10.1210/jcem.76.2.8432797.
- [Background] Yang Y, Zheng S, Li K. [Treatment of uterine leiomyoma by two different doses of mifepristone]. Zhonghua Fu Chan Ke Za Zhi. 1996 Oct;31(10):624-6. Chinese. PMID 9275461
- [Background] Murphy AA, Morales AJ, Kettel LM, Yen SS. Regression of uterine leiomyomata to the antiprogesterone RU486: dose-response effect. Fertil Steril. 1995 Jul;64(1):187-90. PMID 7789557
- [Derived] Yerushalmi GM, Gilboa Y, Jakobson-Setton A, Tadir Y, Goldchmit C, Katz D, Seidman DS. Vaginal mifepristone for the treatment of symptomatic uterine leiomyomata: an open-label study. Fertil Steril. 2014 Feb;101(2):496-500. doi: 10.1016/j.fertnstert.2013.10.015. Epub 2013 Nov 9. PMID 24220703